CLINICAL TRIAL: NCT01864369
Title: Canadian e-Platform to Promote Behavioral Self-Management in Chronic Heart Failure: CHF-CePPORT
Acronym: CHF-CePPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Robert Nolan, Research Psychologist- Director, Behavioral Cardiology Research Unit, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MOP 126118
Record Dates: First submitted 2013-05-15; First posted 2013-05-29 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; e-counseling; quality of life; self-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: eInfo + Usual Care (Active Comparator): Usual Care + eInfo on general guidelines for heart healthy living
  Interventions: Behavioral: eCounseling + Usual Care
- Behavioral: eCounseling + Usual Care (Experimental): Behavioral:eCounseling + Usual Care: interactive web pages utilized to provide e-counseling messages and e-tools.
  Interventions: Behavioral: eCounseling + Usual Care

INTERVENTIONS:
Behavioral: eCounseling + Usual Care — This intervention will use film vignettes and interactive web pages. The e-counseling messages will promote: (i) validation of the subject's stage of "readiness" for behavior change, (ii) collaborative participation by means of subject-selected menus, (iii) reinforcement of "change talk" to resolve ambivalence, (iv) use of self-help information and e-tools for self-monitoring of targeted self-care behaviors, and (v) development of cognitive-behavioral skills to build and strengthen efficacy. Messages will be proactively sent to Controls according to the following schedule: weekly for months 1 to 4, bi-weekly for months 5 to 8, and monthly for months 9 to 12.

SUMMARY:
Chronic Heart Failure (CHF) is a growing public health issue in Canada. Hospital re-admission within 1-year after diagnosis is 25-40%, and the 5-year rate of CHF death is 50%. Counseling by multidisciplinary health care teams helps CHF patients to improve self-care behaviors (for medications, diet, exercise, smoking cessation and symptom monitoring), and this reduces the rate of death and CHF hospitalization. In the absence of intervention, patient adherence to these behaviors is below recommended standards and quality of life among CHF patients becomes progressively compromised. A major challenge is to make self-care counseling available without overtaxing health care resources.

This year multicenter clinical trial will establish and evaluate a Canadian e-platform that provides multidisciplinary e-counseling to help patients with CHF to initiate and maintain recommended self-care behaviors. The investigators will recruit 298 CHF patients in Toronto, Montreal and Vancouver. The investigators hypothesize that a 12-month program of e-Counseling + Usual Care versus general eInfo + Usual Care will improve quality of life, self-care behaviors, program engagement, and heart health. This proposal is based upon previous clinical trials in CHF, e-health and preventive lifestyle counseling by our team. The novel contribution of this research is that it will establish an infrastructure for a pan-Canadian e-platform in preventive e-counseling for CHF. A key feature of this proposal is that our multidisciplinary team will work with professional heart health organizations to share our findings and e-health resources with the public and other health care professionals in Canada, which will help to galvanize research and clinical work in eCounseling. Our clinical trial will strengthen eCounseling services in order to improve the quality of life of patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years of age who are diagnosed with heart failure with reduced ejection fraction ("systolic HF") corresponding to New York Heart Association Class II-III for 3 months prior to enrolment;
2. documentation of LVEF 40%;
3. subject has access to a personal computer;

Exclusion Criteria:

1. Documentation at enrolment of renal failure, significant liver disease or poorly controlled diabetes mellitus;
2. persistent systolic or diastolic hypertension [systolic > 170 mmHg or diastolic > 100 mmHg despite antihypertensive therapy;
3. CHF secondary to cardiovascular co-morbidities/procedures;
4. previous heart transplant or wait listed for heart transplant at time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2013-09; Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life: Kansas City Cardiomyopathy Questionnaire | 12 months
  The primary outcome in CHF-CePPORT is quality of life, as measured by the number of subjects who demonstrate a clinically meaningful increase of ≥5 points on the summary index of the Kansas City Cardiomyopathy Questionnaire (KCCQ).

SECONDARY OUTCOMES:
Program engagement and usability | 4- and 12- months
  Active engagement with digital platform: total time, # logons, % material accessed
Behavioral,functional and clinical outcomes | 4- and 12- months
  Quality of life: number of subjects with KCCQ ≥5 points
Behavioral, clinical and funcitonal outcomes | 4 and 12- months
  Adherence to daily dietary guidelines for fruit and vegetable intake: NIH/NCI Diet History Questionnaire.
Behavioral, functional and clinical outcomes | 4- and 12- months
  Physical activity: 4-day step count with Triaxial Accelerometer.
Behavioral, functional and clinical outcomes | 4- and 12- months
  Self-reported daily activity: The Physical Activity Scale for the Elderly.
Behavioral, functional and clinical outcomes | 4- and 12- months
  Psychological adjustment: Patient Health Questionnaire - 9-item scale (Depression)
Clinical and functional assesments. | 12-months
  Functional capacity: 6-minute walk test.
Behavioral, functional and clinical outcomes | 4- and 12- months
  Patient Health Questionnaire: PHQ-9 (Depression) and GAD-7 (Anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Nolan, PhD, Principal Investigator — University Health Network- University of Toronto
Locations (3):
- Canada (3):
  - St.Paul's Hospital- UBC, Vancouver, British Columbia
  - University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Derived] Nolan RP, Syed F, Stogios N, Maunder R, Sockalingam S, Tai ES, Cobain M, Peiris RG, Huszti E. The evaluation of goal-directed activities to promote well-being and health in heart failure: EUROIA scale. J Patient Rep Outcomes. 2024 Apr 29;8(1):47. doi: 10.1186/s41687-024-00723-x. PMID 38683439
- [Derived] Nolan RP, Ross HJ, Farkouh ME, Huszti E, Chan S, Toma M, D'Antono B, White M, Thomas S, Barr SI, Perreault S, McDonald M, Zieroth S, Isaac D, Wielgosz A, Mielniczuk LM. Automated E-Counseling for Chronic Heart Failure: CHF-CePPORT Trial. Circ Heart Fail. 2021 Jan;14(1):e007073. doi: 10.1161/CIRCHEARTFAILURE.120.007073. Epub 2021 Jan 19. PMID 33464959
- [Derived] Nolan RP, Payne AY, Ross H, White M, D'Antono B, Chan S, Barr SI, Gwadry-Sridhar F, Nigam A, Perreault S, Farkouh M, McDonald M, Goodman J, Thomas S, Zieroth S, Isaac D, Oh P, Rajda M, Chen M, Eysenbach G, Liu S, Zbib A. An Internet-Based Counseling Intervention With Email Reminders that Promotes Self-Care in Adults With Chronic Heart Failure: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2014 Jan 30;3(1):e5. doi: 10.2196/resprot.2957. PMID 24480783
- See also: General contact — http://cardiacehealth.uhnresearch.ca/